CLINICAL TRIAL: NCT02038985
Title: An Evaluation of Fluorescence Imaging + ICG Dye (Firefly) for Use in the Visual Diagnosis of Endometriosis: A Prospective Study
Brief Title: Fluorescence Imaging + ICG Dye for Use in the Visual Diagnosis of Endometriosis
Acronym: FIREFLY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 451140
Record Dates: First submitted 2013-12-30; First posted 2014-01-17 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Endometriosis
Keywords: Endometriosis; Robotic Surgery; Diagnostic Imaging
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- + ICG Dye (Firefly) (Other): Participants will receive ICG Dye
  Interventions: Other: Participants will receive ICG Dye

INTERVENTIONS:
Other: Participants will receive ICG Dye — Participants will receive ICG Dye preoperatively for use in the Visual Diagnosis of Endometriosis

SUMMARY:
The purpose of this study is to evaluate the use of fluorescence imaging + Indocyanine Green (ICG) dye ("Firefly"), compared to standard white light imaging in 2D and 3D, for accurate visual diagnosis of endometriosis during a da Vinci robotically guided endometriosis resection procedure.

DETAILED DESCRIPTION:
Fluorescence imaging has been used for visualization of tissue perfusion in colorectal surgery, detection of pathologic primary and metastatic tumors, and measurement of graft patency in cardiovascular surgery. The da Vinci® Firefly Imaging System, through the use of fluorescence imaging, allows surgeons to view high-resolution near infrared images of blood flow and tissue perfusion in real-time during robotic-assisted surgical procedures, such as during a robotic-assisted endometriosis resection.

Using standard white light imaging, endometriotic lesions can appear red and vascular, white and scarred, black, brown, yellow, or almost any color; atypical implants are clear and can seem like normal tissue. However, there are some published reports demonstrating that the lesions of endometriosis are hypervascular and may be visualized radiographically on the basis of this pathologic feature. Because the individual lesions of endometriosis can vary significantly in their appearance under standard white light, using the hypervascular characteristic of this disease along with the Firefly technology may provide consistency in intraoperative visual diagnosis, and thus may aid the detection and resection of endometriosis.

The ability to accurately visualize all the lesions of endometriosis, typical and atypical in appearance, and thus facilitate complete resection of the disease, may have a significant impact on symptomatic relief and disease recurrence. The Firefly Imaging System of fluorescence imaging + ICG dye may allow for more accurate visual diagnosis of endometriosis during a robotic-assisted endometriosis resection procedure, and therefore may have a positive impact for patients with this disease.

This is a prospective, comparison, single-center, observational study to evaluate fluorescence imaging + ICG dye (Firefly), compared to standard white light imaging in 2D and 3D, for accurate visual diagnosis of endometriosis during a da Vinci endometriosis resection procedure.

ELIGIBILITY:
Inclusion Criteria:

* Be premenopausal (menopause is defined as amenorrhea lasting one year or longer)
* Have symptoms consistent with endometriosis, including the presence of one or more of the following: dysmenorrhea; dyspareunia; chronic pelvic pain (>6 months duration); pressure on the bladder or rectum causing difficult or painful bowel movements; infertility.
* Be willing to undergo planned da Vinci Endometriosis Resection Procedure

Exclusion Criteria:

* Known or suspected allergy to iodine, shellfish, or ICG dye
* Presence of medical conditions contraindicating general anesthesia or standard laparoscopic/ robotic surgery
* Active pelvic infection
* Previous history of radiation therapy to the pelvis
* Known or suspected pregnancy
* Presence of anatomy unsuitable for laparoscopic surgery
* Previously undiagnosed intra-abdominal or pelvic malignancy
* Inability of patient to tolerate Trendelenberg position or pneumoperitoneum

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-08-16 (Actual)

PRIMARY OUTCOMES:
Quality of fluorescence imaging using + ICG dye (Firefly). | 1 hour
  Quality is defined by the investigators perception of accuracy of visual diagnosis and how clear are the the resultant images used for visualization and mapping of lesions. The quality of the fluorescence imaging + ICG dye (Firefly) will be compared to standard white light imaging in 2D and 3D for accurate visual diagnosis of endometriosis during a da Vinci endometriosis resection procedure

SECONDARY OUTCOMES:
Quality of Life | 3 months
  Quality of Life (QOL) will be captured by utilizing the validated questionnaire SF-36 short form, administered at three time-points: pre-operative, at 3-months post-operative, and at 6-months post-operative. The QOL aspects examined with the SF-36 include vitality, mental health physical functioning, bodily pain, general health perceptions, as well as physical, emotional, and social role functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Aileen Caceres, MD, Principal Investigator — Florida Hospital Celebration Health
Locations (1):
- Florida Hospital Celebration Health, Celebration, Florida, United States